CLINICAL TRIAL: NCT01596647
Title: A Phase I, Multi-center, Open-label, Drug-drug Interaction Study to Assess the Effect of TKI258 on the Pharmacokinetics of Caffeine, Diclofenac, Omeprazole and Midazolam Administered as a Four-drug Cocktail in Patients With Advanced Solid Tumors, Excluding Breast Cancer
Brief Title: Pharmacokinetic Drug-drug Interaction Study of Dovitinib (TKI258) in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTKI258A2119; 2011-001489-16 (EudraCT Number)
Record Dates: First submitted 2012-03-23; First posted 2012-05-11 (Estimated); Last update posted 2020-12-21 (Actual); Status verified 2015-05

CONDITIONS: Advanced Solid Tumors, Excluding Breast Cancer
Keywords: cancer, tumors, phase I, drug-drug interaction, pharmacokinetic, probe drug, caffeine, diclofenac, omeprazole, midazolam, CYP1A2, CYP2C9, CYP2C19, CYP3A4
MeSH Terms: conditions — Neoplasms | interventions — Caffeine; Diclofenac; Omeprazole; Midazolam; 4-amino-5-fluoro-3-(5-(4-methylpiperazin-1-yl)-1H-benzimidazol-2-yl)quinolin-2(1H)-one

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- TKI258 (dovitinib) (Experimental): dovitinib, 5 days on / 2 days off dose schedule
  Interventions: Drug: caffeine; Drug: diclofenac; Drug: omeprazole; Drug: midazolam; Drug: TKI258

INTERVENTIONS:
Drug: caffeine — single dose of the probe drug cocktail contains: caffeine, diclofenac, omeprazole and midazolam
  Other Names: probe drug
Drug: diclofenac — single dose of the probe drug cocktail contains: caffeine, diclofenac, omeprazole and midazolam
  Other Names: probe drug
Drug: omeprazole — single dose of the probe drug cocktail contains: caffeine, diclofenac, omeprazole and midazolam
  Other Names: probe drug
Drug: midazolam — single dose of the probe drug cocktail contains: caffeine, diclofenac, omeprazole and midazolam
  Other Names: probe drug
Drug: TKI258 — dovitinib, 5 days on / 2 days off dose schedule
  Other Names: dovitinib

SUMMARY:
This is a multi-center, open-label, phase I study to assess the effects of dovitinib (TKI258) on the pharmacokinetics of a cocktail of caffeine, diclofenac, omeprazole and midazolam in patients with advanced solid tumors, excluding breast cancer. The aim of this study is to evaluate the potential effect of dovitinib (TKI258) on the metabolism of the probe drugs caffeine, diclofenac, omeprazole and midazolam, which are metabolized by CYP1A2, CYP2C9, CYP2C19 and CYP3A4 respectively (Cytochrome P450 isoenzyme), comparing the single-dose pharmacokinetics (AUCtlast, AUCinf and Cmax parameters) of each of the individual probe drug co-administered with and without multiple dose of dovitinib (TKI258) 500 mg under a 5 days on / 2 days off dose schedule. The study foresees two treatment phases: DDI (drug-drug interaction) followed by post-DDI. During the DDI phase patients receive treatment with the probe drug cocktail and dovitinib (TKI258). During the post-DDI phase patients may continue to receive treatment with dovitinib (TKI258) until disease progression (assessed by RECIST 1.1), unacceptable toxicity, death or discontinuation from the study treatment for any other reason.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a cytopathologically or histopathologically confirmed diagnosis of an advanced solid tumor, excluding breast cancer which has progressed despite standard therapy or for which no standard therapy exists
* ECOG performance status 0 or 1 and anticipated life expectancy ≥ 3 months
* Patient must meet protocol-specific laboratory values

Exclusion Criteria:

* Patients with brain metastases
* Patients who have received or who are expected to receive any prohibited medications and therapies
* Patients who have received CYP1A2 inducer, CYP2C9/2C19 inducer or CYP3A4 inducer medications within 30 days prior to start study treatment or are expected to receive during the first 14 days after starting the study treatment
* Patients with a known hypersensitivity to benzodiazepines
* Patients who have not recovered from previous anti-cancer therapies
* Patient with impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of TKI258
* Patients who have concurrent severe and/or uncontrolled concomitant medical conditions that could compromise participation in the study
* Female patients who are pregnant or breast-feeding
* Fertile males or women not willing to use highly effective methods of contraception
* Other protocol-defined inclusion/exclusion criteria will apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-05; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Probe substrate pharmacokinetics (PK) parameters: Cmax (Maximum (peak) concentration of drug) | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),
Probe substrate PK parameters: AUCtlast (Area Under the Curve) | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),
Probe substrate PK parameters: AUCinf | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),
Probe substrate PK parameters:Tmax (Time to maximum concentration) | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),
Probe substrate PK parameters: HL (Half-life time) | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),
Probe substrate PK parameters:CL/F (Apparent Oral Clearance) | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),
Probe substrate PK parameters:Vz/F (apparent volume of distribution) | multiple time-points over 24h post dose on day 1 and Day 13 (DDI phase),

SECONDARY OUTCOMES:
Frequency and severity of AEs (Adverse Events) | up to at least 30 days after the last dose of dovitinib (TKI258)
Preliminary evidence of antitumor activity of dovitinib (TKI258) | every 8 weeks until progression of disease
  overall response based on investigator's assessment and best overall response using RECIST 1.1
Frequency and severity of SAEs (Serious Adverse Events) | up to at least 30 days after the last dose of dovitinib (TKI258)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (5):
- United States (5):
  - University of Kansas Cancer Center Medical Center, Kansas City, Kansas
  - Henry Ford Hospital Henry Ford, Detroit, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Comprehensive Cancer Centers, Las Vegas, Nevada
  - Cancer Institute of New Jersey Dept of Cancer Institute of NJ, New Brunswick, New Jersey

REFERENCES:
- See also: Results for CTKI258A2119 can be found on the Novartis Clinical Trial Results Website — https://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=13883